CLINICAL TRIAL: NCT00768898
Title: Defining the Conjunctival Staining Method: Instillation Volume and Time Course to Assess Staining With Lissamine Green
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: M-08-01
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Conjunctival Staining
Keywords: conjunctival; staining

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2.5 microliters lissamine green
  Interventions: Other: 2.5/5.0/10.0 ÂµL lissamine green
- 5.0 microliters lissamine green
  Interventions: Other: 2.5/5.0/10.0 ÂµL lissamine green
- 10.0 microliters lissamine green
  Interventions: Other: 2.5/5.0/10.0 ÂµL lissamine green

INTERVENTIONS:
Other: 2.5/5.0/10.0 ÂµL lissamine green — vital stain solution

SUMMARY:
The purpose of this study is to determine the correct volume of lissamine green to use when assessing conjunctival staining, and to determine the time course needed to evaluate conjunctival staining after lissamine green has been instilled in the eye.

ELIGIBILITY:
Inclusion Criteria:

* conjunctival staining

Exclusion Criteria:

* ocular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 subjects with conjunctival staining and no other ocular pathology were recruited and enrolled.
Pre-assignment Details: This reporting group includes all enrolled participants.
Groups:
- Overall: All enrolled participants
Period: Overall Study
Arm/Group | Overall
Started | 30
Completed | 28
Not Completed | 2
Not completed — Unrelated injury | 1
Not completed — Headache | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Staining at 1 Minute
Description: Lissamine green was instilled in each eye. Conjunctival staining was assessed by the investigator in the nasal and temporal sections. The Oxford Scheme was used for each section, with a possible score of 0-5 for each section, where 0=absent and 5=severe. The nasal and temporal scores were summed, for a possible score of 0-10 for each eye. Each subject was represented by a single eye, referred to as the "study eye." The study eye was defined as the eye that attained the highest stain at any measurement time point during the screening visit.
Time Frame: 1 minute after instillation
Population: Analysis conducted per protocol. All subjects participated in each arm/group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 2.5 Microliters Lissamine Green: 2.5 microliters lissamine green were instilled in each eye.
- 5.0 Microliters Lissamine Green: 5.0 microliters lissamine green instilled in each eye
- 10.0 Microliters Lissamine Green: 10.0 microliters lissamine green instilled in each eye
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Number analyzed (Participants) | 21 | 21 | 21
Units on a scale | 3.29 (1.58) | 3.67 (1.72) | 3.98 (1.75)

2. Primary Outcome: Conjunctival Staining at 2 Minutes
Description: as for outcome 1
Time Frame: 2 minutes after instillation
Population: Analysis conducted per protocol. All subjects participated in each arm/group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 2.5 Microliters Lissamine Green: 2.5 microliters lissamine green instilled in each eye
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Number analyzed (Participants) | 21 | 21 | 21
Units on a scale | 3.67 (1.75) | 4.29 (1.76) | 4.64 (1.75)

3. Primary Outcome: Conjunctival Staining at 3 Minutes
Description: as for outcome 1
Time Frame: 3 minutes after instillation
Population: Analysis conducted per protocol. All subjects participated in each arm/group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Number analyzed (Participants) | 21 | 21 | 21
Units on a scale | 3.02 (1.60) | 3.88 (1.85) | 4.12 (1.92)

4. Primary Outcome: Conjunctival Staining at 4 Minutes
Description: as for outcome 1
Time Frame: 4 minutes after instillation
Population: Analysis conducted per protocol. All subjects participated in each arm/group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Number analyzed (Participants) | 21 | 21 | 21
Units on a scale | 2.48 (1.63) | 3.14 (1.75) | 3.69 (1.81)

5. Primary Outcome: Conjunctival Staining at 5 Minutes
Description: as for outcome 1
Time Frame: 5 minutes after instillation
Population: Analysis conducted per protocol. All subjects participated in each arm/group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Number analyzed (Participants) | 21 | 21 | 21
Units on a scale | 2.12 (1.48) | 2.67 (1.78) | 3.10 (1.64)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Groups:
- 2.5 Microliters Lissamine Green: 2.5 microliters lissamine green
- 5.0 Microliters Lissamine Green: 5.0 microliters lissamine green
- 10.0 Microliters Lissamine Green: 10.0 microliters lissamine green
Arm/Group | 2.5 Microliters Lissamine Green | 5.0 Microliters Lissamine Green | 10.0 Microliters Lissamine Green
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes